CLINICAL TRIAL: NCT00389220
Title: A Randomized Comparison of a Biolimus-Eluting Stent With a Sirolimus-Eluting Stent for Percutaneous Coronary Intervention
Brief Title: Limus Eluted From A Durable Versus ERodable Stent Coating
Acronym: LEADERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05EU01
Record Dates: First submitted 2006-10-13; First posted 2006-10-18 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Coronary Disease; Coronary Stenosis
Keywords: Coronary Disease; Coronary Stenosis; Angioplasty; Coronary Restenosis; Drug Eluting Stent
MeSH Terms: conditions — Coronary Disease; Coronary Stenosis; Coronary Restenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BioMatrix Flex stent (Active Comparator): Coronary stent placement with Biolimus A9 coated stent with biodegradable polymer
  Interventions: Device: Coronary stent placement
- Cypher Select stent (Active Comparator): Coronary stent placement with Sirolimus coated stent with durable polymer
  Interventions: Device: Coronary stent placement

INTERVENTIONS:
Device: Coronary stent placement — Coronary stent placement

SUMMARY:
The purpose of this study is to compare the BioMatrix Flex (Biolimus A9-Eluting) stent system with the Cypher SELECT (Sirolimus-Eluting) stent system in a non-inferiority trial.

DETAILED DESCRIPTION:
Compare the safety and efficacy of the BioMatrix Flex (Biolimus A9-Eluting) stent system with the Cypher SELECT (Sirolimus-Eluting) stent system in a prospective, multi-center, randomized, controlled, non-inferiority trial in patients undergoing percutaneous coronary intervention in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes including non-ST elevation myocardial infarction and ST-elevation myocardial infarction;
* Presence of one or more coronary artery stenoses >50% in a native coronary artery or a saphenous bypass graft from 2.25 to 3.5 mm in diameter that can be covered with one or multiple stents;
* No limitation on the number of treated lesions, and vessels, and lesion length

Exclusion Criteria:

* Pregnancy;
* Known intolerance to aspirin, clopidogrel, heparin, stainless steel, Sirolimus, Biolimus or contrast material;
* Inability to provide informed consent;
* Currently participating in another trial before reaching first endpoint;
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the perisurgical period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1707 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 9 month
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 30 days
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
Cardiac death | 30 days
  Cardiac death
All deaths | 30 days
  All deaths (cardiac and non-cardiac)
Myocardial infarction | 30 days
  Myocardial infarction (Q-wave and NQWMI)
Angiographic and clinical stent thrombosis. | 30 days
  Angiographic and clinical stent thrombosis
In-stent and in-segment binary restenosis rate as assessed by QCA. | 9 month
  In-stent and in-segment binary restenosis rate as assessed by QCA.
In-stent and in-segment minimal luminal diameter (MLD) as assessed by QCA. | 9 month
  In-stent and in-segment minimal luminal diameter (MLD) as assessed by QCA
In-segment percent diameter stenosis (%DS). | 9 month
  In-segment percent diameter stenosis (%DS) as assessed by QCA
In-stent and in-segment late luminal loss | 9 month
  In-stent and in-segment late luminal loss as assessed by QCA
Device success, lesion success and procedural success. | at implant
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 6 month
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 1 year
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 2 years
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
Cardiac death | 6 month
  Cardiac death
Cardiac death | 9 month
  Cardiac death
Cardiac death | 1 year
  Cardiac death
Cardiac death | 2 year
  Cardiac death
Cardiac death | 3 year
  Cardiac death
Cardiac death | 4 year
  Cardiac death
Cardiac death | 5 year
  Cardiac death
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 3 year
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 4 year
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
Major adverse cardiac events (MACE) in the overall population according to the ARC definitions. | 5 year
  Major adverse cardiac events (MACE) in the overall population defined as composite of cardiac death,myocardial infarction (Q-wave and Non-Q wave)justified target vessel revascularization and Justified and non-justified target lesion revascularization (TLR)
All deaths | 6 month
  All deaths (cardiac and non-cardiac)
All deaths | 9 month
  All deaths (cardiac and non-cardiac)
All deaths | 1 year
  All deaths (cardiac and non-cardiac)
All deaths | 2 years
  All deaths (cardiac and non-cardiac)
All deaths | 3 years
  All deaths (cardiac and non-cardiac)
All deaths | 4 years
  All deaths (cardiac and non-cardiac)
All deaths | 5 years
  All deaths (cardiac and non-cardiac)
Myocardial infarction | 6 month
  Myocardial infarction (Q-wave and NQWMI)
Myocardial infarction | 9 month
  Myocardial infarction (Q-wave and NQWMI)
Myocardial infarction | 1 year
  Myocardial infarction (Q-wave and NQWMI)
Myocardial infarction | 2 years
  Myocardial infarction (Q-wave and NQWMI)
Myocardial infarction | 3 years
  Myocardial infarction (Q-wave and NQWMI)
Myocardial infarction | 4 years
  Myocardial infarction (Q-wave and NQWMI)
Myocardial infarction | 5 years
  Myocardial infarction (Q-wave and NQWMI)
Angiographic and clinical stent thrombosis. | 6 month
  Angiographic and clinical stent thrombosis
Angiographic and clinical stent thrombosis. | 9 month
  Angiographic and clinical stent thrombosis
Angiographic and clinical stent thrombosis. | 1 year
  Angiographic and clinical stent thrombosis
Angiographic and clinical stent thrombosis. | 2 years
  Angiographic and clinical stent thrombosis
Angiographic and clinical stent thrombosis. | 3 years
  Angiographic and clinical stent thrombosis
Angiographic and clinical stent thrombosis. | 4 years
  Angiographic and clinical stent thrombosis
Angiographic and clinical stent thrombosis. | 5 years
  Angiographic and clinical stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, Prof., Principal Investigator — Medizinische Universitätsklinik, Swiss Cardiovacular Center Bern
Locations (10):
- Onze Lieve Vrouw Ziekenhuis, Cardiologisch Centrum, Moorselbaan 164, Aalst, Belgium
- L'Institut Cardiovasculaire Paris Sud, Institut Hospitalier Jacques Cartier, Service de Coronarographie, 6, Avenue du Noyer Lambert, Massy, France
- Germany (3):
  - Herzzentrum Leipzig, Innere Medizin/Kardiologie, Struimpellstrasse 39, Leipzig
  - Universitatsklinikum Munchen, Medizinische Klinik Kardiologie, Ziemssenstrasse 1, Munich
  - Klinikum Bogenhausen der Stad München, Abteilung für Kardiologie und Pnemlogie, Englschalkstrasse 77, Munich
- University Medical Center Rotterdam Erasmus, Thoraxcentrum, Rotterdam, Netherlands
- American Heart of Poland Sp. z o.o., Dąbrowa Górnicza, Poland
- Switzerland (2):
  - Medizinische Universitätsklinik, Swiss Cardiovacular Center Bern, Inselspital, Bern
  - University Hospital Zürich, Director of Invasive Cardiology, Rämistrasse 100, Zurich
- Royal Brompton Hospital, Sydney Street, London, United Kingdom

REFERENCES:
- [Result] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Result] Garg S, Sarno G, Serruys PW, de Vries T, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, Di Mario C, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P, Windecker S. The twelve-month outcomes of a biolimus eluting stent with a biodegradable polymer compared with a sirolimus eluting stent with a durable polymer. EuroIntervention. 2010 Jun;6(2):233-9. PMID 20562074
- [Result] Sarno G, Garg S, Onuma Y, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, van Geuns RJ, Eerdmans P, Garcia-Garcia HM, van Es GA, Goedhart D, de Vries T, Juni P, Meier B, Windecker S, Serruys P. The impact of body mass index on the one year outcomes of patients treated by percutaneous coronary intervention with Biolimus- and Sirolimus-eluting stents (from the LEADERS Trial). Am J Cardiol. 2010 Feb 15;105(4):475-9. doi: 10.1016/j.amjcard.2009.09.055. Epub 2010 Jan 5. PMID 20152241
- [Result] Wykrzykowska JJ, Serruys PW, Onuma Y, de Vries T, van Es GA, Buszman P, Linke A, Ischinger T, Klauss V, Corti R, Eberli F, Wijns W, Morice MC, di Mario C, van Geuns RJ, Juni P, Windecker S. Impact of vessel size on angiographic and clinical outcomes of revascularization with biolimus-eluting stent with biodegradable polymer and sirolimus-eluting stent with durable polymer the LEADERS trial substudy. JACC Cardiovasc Interv. 2009 Sep;2(9):861-70. doi: 10.1016/j.jcin.2009.05.024. PMID 19778775
- [Result] Wykrzykowska JJ, Raber L, de Vries T, Bressers M, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Regar E, Juni P, Windecker S, Serruys PW. Biolimus-eluting biodegradable polymer versus sirolimus-eluting permanent polymer stent performance in long lesions: results from the LEADERS multicentre trial substudy. EuroIntervention. 2009 Aug;5(3):310-7. doi: 10.4244/v5i3a49. PMID 19736154
- [Derived] Yuan H, Wu Z, Lu T, Wei T, Zeng Y, Liu Y, Huang C. Comparison of biodegradable and durable polymer drug-eluting stents in acute coronary syndrome: a meta-analysis. BMJ Open. 2022 Jun 8;12(6):e058075. doi: 10.1136/bmjopen-2021-058075. PMID 35676012
- [Derived] Koskinas KC, Siontis GC, Piccolo R, Franzone A, Haynes A, Rat-Wirtzler J, Silber S, Serruys PW, Pilgrim T, Raber L, Heg D, Juni P, Windecker S. Impact of Diabetic Status on Outcomes After Revascularization With Drug-Eluting Stents in Relation to Coronary Artery Disease Complexity: Patient-Level Pooled Analysis of 6081 Patients. Circ Cardiovasc Interv. 2016 Feb;9(2):e003255. doi: 10.1161/CIRCINTERVENTIONS.115.003255. PMID 26823484
- [Derived] Grundeken MJ, Wykrzykowska JJ, Ishibashi Y, Garg S, de Vries T, Garcia-Garcia HM, Onuma Y, de Winter RJ, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Meier B, Juni P, Yazdani A, Copt S, Windecker S, Serruys PW. First generation versus second generation drug-eluting stents for the treatment of bifurcations: 5-year follow-up of the LEADERS all-comers randomized trial. Catheter Cardiovasc Interv. 2016 Jun;87(7):E248-60. doi: 10.1002/ccd.26344. Epub 2015 Dec 9. PMID 26649651
- [Derived] Zhang YJ, Iqbal J, Windecker S, Linke A, Antoni D, Sohn HY, Corti R, van Es GA, Copt S, Eerdmans P, Saitta R, Morice MC, Di Mario C, Juni P, Wijns W, Buszman P, Serruys PW. Biolimus-eluting stent with biodegradable polymer improves clinical outcomes in patients with acute myocardial infarction. Heart. 2015 Feb;101(4):271-8. doi: 10.1136/heartjnl-2014-306359. Epub 2014 Nov 25. PMID 25423953
- [Derived] Vranckx P, Kalesan B, Stefanini GG, Farooq V, Onuma Y, Silber S, de Vries T, Juni P, Serruys PW, Windecker S. Clinical outcome of patients with stable ischaemic heart disease as compared to those with acute coronary syndromes after percutaneous coronary intervention. EuroIntervention. 2015 Jun;11(2):171-9. doi: 10.4244/EIJV11I2A31. PMID 24531331
- [Derived] Serruys PW, Farooq V, Kalesan B, de Vries T, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Wijns W, Morice MC, Di Mario C, Corti R, Antoni D, Sohn HY, Eerdmans P, Rademaker-Havinga T, van Es GA, Meier B, Juni P, Windecker S. Improved safety and reduction in stent thrombosis associated with biodegradable polymer-based biolimus-eluting stents versus durable polymer-based sirolimus-eluting stents in patients with coronary artery disease: final 5-year report of the LEADERS (Limus Eluted From A Durable Versus ERodable Stent Coating) randomized, noninferiority trial. JACC Cardiovasc Interv. 2013 Aug;6(8):777-89. doi: 10.1016/j.jcin.2013.04.011. PMID 23968698
- [Derived] Gutierrez-Chico JL, Raber L, Regar E, Okamura T, di Mario C, van Es GA, Windecker S, Serruys PW. Tissue coverage and neointimal hyperplasia in overlap versus nonoverlap segments of drug-eluting stents 9 to 13 months after implantation: in vivo assessment with optical coherence tomography. Am Heart J. 2013 Jul;166(1):83-94. doi: 10.1016/j.ahj.2013.04.001. Epub 2013 May 3. PMID 23816026
- [Derived] Stefanini GG, Kalesan B, Pilgrim T, Raber L, Onuma Y, Silber S, Serruys PW, Meier B, Juni P, Windecker S. Impact of sex on clinical and angiographic outcomes among patients undergoing revascularization with drug-eluting stents. JACC Cardiovasc Interv. 2012 Mar;5(3):301-10. doi: 10.1016/j.jcin.2011.11.011. PMID 22440496
- [Derived] Gutierrez-Chico JL, Juni P, Garcia-Garcia HM, Regar E, Nuesch E, Borgia F, van der Giessen WJ, Davies S, van Geuns RJ, Secco GG, Meis S, Windecker S, Serruys PW, di Mario C. Long-term tissue coverage of a biodegradable polylactide polymer-coated biolimus-eluting stent: comparative sequential assessment with optical coherence tomography until complete resorption of the polymer. Am Heart J. 2011 Nov;162(5):922-31. doi: 10.1016/j.ahj.2011.09.005. Epub 2011 Oct 7. PMID 22093210
- [Derived] Stefanini GG, Kalesan B, Serruys PW, Heg D, Buszman P, Linke A, Ischinger T, Klauss V, Eberli F, Wijns W, Morice MC, Di Mario C, Corti R, Antoni D, Sohn HY, Eerdmans P, van Es GA, Meier B, Windecker S, Juni P. Long-term clinical outcomes of biodegradable polymer biolimus-eluting stents versus durable polymer sirolimus-eluting stents in patients with coronary artery disease (LEADERS): 4 year follow-up of a randomised non-inferiority trial. Lancet. 2011 Dec 3;378(9807):1940-8. doi: 10.1016/S0140-6736(11)61672-3. Epub 2011 Nov 8. PMID 22075451
- [Derived] Klauss V, Serruys PW, Pilgrim T, Buszman P, Linke A, Ischinger T, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, van Geuns RJ, van Es GA, Kalesan B, Wenaweser P, Juni P, Windecker S. 2-year clinical follow-up from the randomized comparison of biolimus-eluting stents with biodegradable polymer and sirolimus-eluting stents with durable polymer in routine clinical practice. JACC Cardiovasc Interv. 2011 Aug;4(8):887-95. doi: 10.1016/j.jcin.2011.03.017. PMID 21851904
- [Derived] Gutierrez-Chico JL, Regar E, Nuesch E, Okamura T, Wykrzykowska J, di Mario C, Windecker S, van Es GA, Gobbens P, Juni P, Serruys PW. Delayed coverage in malapposed and side-branch struts with respect to well-apposed struts in drug-eluting stents: in vivo assessment with optical coherence tomography. Circulation. 2011 Aug 2;124(5):612-23. doi: 10.1161/CIRCULATIONAHA.110.014514. Epub 2011 Jul 18. PMID 21768536
- [Derived] Wykrzykowska JJ, Garg S, Onuma Y, de Vries T, Goedhart D, Morel MA, van Es GA, Buszman P, Linke A, Ischinger T, Klauss V, Corti R, Eberli F, Wijns W, Morice MC, di Mario C, van Geuns RJ, Juni P, Windecker S, Serruys PW. Value of age, creatinine, and ejection fraction (ACEF score) in assessing risk in patients undergoing percutaneous coronary interventions in the 'All-Comers' LEADERS trial. Circ Cardiovasc Interv. 2011 Feb 1;4(1):47-56. doi: 10.1161/CIRCINTERVENTIONS.110.958389. Epub 2011 Jan 4. PMID 21205944
- [Derived] Wykrzykowska JJ, Garg S, Girasis C, de Vries T, Morel MA, van Es GA, Buszman P, Linke A, Ischinger T, Klauss V, Corti R, Eberli F, Wijns W, Morice MC, di Mario C, van Geuns RJ, Juni P, Windecker S, Serruys PW. Value of the SYNTAX score for risk assessment in the all-comers population of the randomized multicenter LEADERS (Limus Eluted from A Durable versus ERodable Stent coating) trial. J Am Coll Cardiol. 2010 Jul 20;56(4):272-7. doi: 10.1016/j.jacc.2010.03.044. PMID 20633818